CLINICAL TRIAL: NCT00782613
Title: Randomized, Double-Blind, Placebo-Controlled Study of Efficacy and Wafety of Topical ALT-2074 (SYI-2074) for Treatment of Chronic
Brief Title: Efficacy and Safety of Topical ALT-2074 (SYI-2074) for Treatment of Chronic Plaque Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been termination early due to financial contraints.
Sponsor: Synvista Therapeutics, Inc (Industry)
Responsible Party: Moshe Neuman Ph.D., Biomedical Research Design, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-2074-205; NCT00757861 (obsolete NCT alias)
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; The primary objective of this study will be to evaluate the; efficacy of topical ALT-2074 applied twice daily for 28; days for treatment of chronic plaque psoriasis in adult; subjects.; The secondary objective will be to evaluate the safety; of topical ALT-2074 applied twice daily for 28 days for; treatment of chronic plaque psoriasis in adult subjects.; Tertiary objectives will be to provide visual documentation; of the improvement of psoriatic plaques treated with; ALT-2074 using digital photography, and to determine the; extent of systemic absorption of topically applied ALT-2074; based on a pharmacokinetic measurement of blood; concentration.
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Two psoriatic plaques of similar surface area and severity will be identified for each subject. ALT-2074 will be applied topically twice daily to 1 of the 2 target plaques, and the placebo control to the other plaque for a period of 28 days in amounts sufficient to cover the entire surface area of the target plaque, extending to 1 cm outside of the plaque border.
  Interventions: Drug: 4,4-dimethyl-benziso-2H-selenazine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4,4-dimethyl-benziso-2H-selenazine — ALT-2074 in a 0.5% cream formulation
  Arms: 1
Drug: Placebo — Placebo in a cream formulation
  Arms: 2

SUMMARY:
The primary objective of this study will be to evaluate the efficacy of topical ALT-2074 applied twice daily for 28 days for treatment of chronic plaque psoriasis in adult subjects.

The secondary objective will be to evaluate the safety of topical ALT-2074 applied twice daily for 28 days for treatment of chronic plaque psoriasis in adult subjects.

Tertiary objectives will be to provide visual documentation of the improvement of psoriatic plaques treated with ALT-2074 using digital photography, and to determine the extent of systemic absorption of topically applied ALT-2074 based on a pharmacokinetic measurement of blood concentration.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to qualify for entry into the study:

1. Men and women between 18 and 75 years old, inclusive.
2. Clinical diagnosis of stable, chronic plaque psoriasis for at least 6 months prior to Visit 1.
3. In otherwise good general health and free of any disease or physical condition which might impair evaluation of plaque psoriasis.
4. Plaque psoriasis treatable area <10% BSA. (Subject palm size is equivalent to 1% of BSA.)
5. Have 2 well-matched plaques (target plaques) of approximately 3 to 8 cm by 3 to 8 cm in size in areas on the right and left or front and back, at sites other than the knees, below the knees, elbows, head, face, scalp, palms, and intertriginous areas.
6. A Combined Psoriasis Severity Score (CPSS) > 6 for each target plaque at Visit 1.
7. Willing to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
8. Able to understand and willing to comply with all study requirements, particularly the regimen for administration of study drug.
9. Able to understand and willing to sign the Informed Consent Form.

Exclusion Criteria:

Any subject who meets any of the following criteria will not qualify for entry into the study:

1. Women who are pregnant, lactating, planning to become pregnant, or women of child-bearing potential who have not successfully been using the same medically acceptable contraceptive methods over the previous 3 months, eg, oral contraceptive agents, intrauterine device (IUD), and barrier method plus spermicide.
2. Clinical diagnosis of guttate, pustular, erythrodermic, or other non-plaque forms of psoriasis.
3. Use of emollients or moisturizers on areas to be treated within 24 hours prior to Visits 1 or 2.
4. Use of topical antipsoriatic therapy (including topical retinoids, corticosteroids, or vitamin D analogs) on the areas to be treated within 2 weeks prior to Visit 2.
5. Received systemic immunomodulatory therapy to treat psoriasis (eg, methotrexate, cyclosporine, alefacept, etanercept, infliximab, efalizumab, adalimumab) within 12 weeks prior to Visit 2.
6. Received phototherapy (including laser), photochemotherapy, or systemic psoriasis therapy (eg, systemic corticosteroids, retinoids such as acitretin) within 4 weeks prior to Visit 2.
7. Recent history (within past 12 months) of alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 4 oz wine, or 1.5 oz distilled spirits).
8. History of noncompliance to medical regimens or unwilling to comply with the study protocol.
9. Participation in an investigational drug study within 30 days prior to Visit 2.
10. Serious or unstable medical or psychological conditions that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of topical ALT-2074 applied twice daily for 28 days for treatment of chronic plaque psoriasis in adult subjects. | 28 days

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Ha'emek Medical Center, Afula
  - Kaplan Medical Center, Rehovot
  - Chaim Sheba Medical Center, Tel Litwinsky